CLINICAL TRIAL: NCT00408005
Title: Intensified Methotrexate, Nelarabine (Compound 506U78) and Augmented BFM Therapy for Children and Young Adults With Newly Diagnosed T-cell Acute Lymphoblastic Leukemia (ALL) or T-cell Lymphoblastic Lymphoma
Brief Title: Combination Chemotherapy in Treating Young Patients With Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00307; NCI-2009-00307 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AALL0434; 07-169; CDR0000514500; AALL0434 (Other: Children's Oncology Group); AALL0434 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: T Acute Lymphoblastic Leukemia; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Leyk; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; nelarabine; pegaspargase; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Thioguanine; Vincristine

ARMS (17):
- Group 0 Induction Therapy (Experimental): All patients (T-ALL and T-LLy) receive cytarabine intrathecally (IT) on day 1; vincristine sulfate IV on days 1, 8, 15, and 22; prednisone IV or PO twice daily BID on days 1-28; pegaspargase IM (may give IV over 1 to 2 hours) on day 4, 5, or 6; daunorubicin hydrochloride IV on days 1, 8, 15 and 22; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease).
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Drug: Vincristine Sulfate
- Group 1 Arm IV (Consolidation chemotherapy) (Active Comparator): Patients receive nelarabine IV over 60 minutes on days 1-5 and 43-47; methotrexate IT on days 15, 22, 57, and 64; cyclophosphamide IV over 30 minutes on days 8 and 50; cytarabine IV over 15-30 minutes or SC on days 8-11, 15-18, 50-53 and 57-60; mercaptopurine PO on days 8-21 and 50-63; vincristine sulfate IV on days 22, 29, 64, and 71; and pegaspargase IM or IV over 1-2 hours on days 22 and 64. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 15, 22-26, and 29-33 (DS patients excluded as of 09/29/10). (Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT QD on days 22-28 and 29-35.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Nelarabine; Drug: Pegaspargase; Radiation: Radiation Therapy
- Group I Arm I (Consolidation chemotherapy) (Active Comparator): Patients receive methotrexate IT on days 1, 8, 15, and 22; cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine IV over 15-30 minutes or SC on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO on days 1-14 and 29-42; vincristine sulfate IV on days 15, 22, 43 and 50; and pegaspargase IM or IV over 1-2 hours on days 15 and 43. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 11-12, 15-19, and 22-26. (DS patients excluded as of 09/29/10.) Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT (1,200 cGy/dose) QD on days 15-21 and 22-28. Patients with low-risk disease do not undergo CRT. Patients with standard risk T-LLy received Arm I, and those with high risk T-LLy were randomized between Arm I and Arm II combination chemotherapy.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Group I Arm I (Delayed intensification chemotherapy (Active Comparator): Patients receive vincristine sulfate IV on days 1, 8, 15, 43, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age and for patients with DS); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6, AND day 43; methotrexate IT on days 1, 29, and 36; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 15-30 minutes or SC on days 29-32 and 36-39; and thioguanine PO on days 29-42. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose (DS patients excluded as of 09/29/10). Standard risk T-LLy patients were assigned to Arm I and those with high risk were randomized between Arm I and Arm II.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group I Arm I (Maintenance chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV on days 1, 29, and 57; prednisone PO BID on days 1-5, 29-33, and 57-61; mercaptopurine PO QD on days 1-84; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; and methotrexate IT on day 1. Treatment repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 119) (for girls with T-ALL), all patients with T-LLy, and 3 years from the start of interim maintenance therapy (approximately week 171) (for boys with T-ALL).
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Prednisone; Drug: Vincristine Sulfate
- Group I Arm I (Interim maintenance chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV and escalating doses of methotrexate IV on days 1, 11, 21, 31, and 41; pegaspargase* IM or IV over 1-2 hours on days 2 and 22; and methotrexate IT on days 1 and 31. Patients with DS also receive leucovorin calcium PO 48 and 60 hours after each methotrexate IT dose (DS patients excluded as of 09/29/10).
  Note: *Patients with an allergy to pegaspargase receive Erwinia asparaginase on days 2, 4, 6, 8, 10, 12, 22, 24, 26, 28, 30, and 32.
  Interventions: Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine Sulfate
- Group I Arm II (Consolidation chemotherapy) (Active Comparator): Patients receive nelarabine IV over 60 minutes on days 1-5 and 43-47; methotrexate IT on days 15, 22, 57, and 64; cyclophosphamide IV over 30 minutes on days 8 and 50; cytarabine IV over 15-30 minutes or SC on days 8-11, 15-18, 50-53 and 57-60; mercaptopurine PO on days 8-21 and 50-63; vincristine sulfate IV on days 22, 29, 64, and 71; and pegaspargase IM or IV over 1-2 hours on days 22 and 64. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 15, 22-26, and 29-33 (DS patients excluded as of 09/29/10). (Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT QD on days 22-28 and 29-35. Patients with high risk T-LLy were either randomized to Arm I or Arm II. Patients with T-LLy who failed induction therapy were assigned to Arm II.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Nelarabine; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Group I Arm II (Delayed intensification chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV on days 1, 8, 15, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6 AND day 50; methotrexate IT on days 1, 36, and 43; nelarabine IV over 60 minutes on days 29-33; cyclophosphamide IV over 30 minutes on day 36; cytarabine IV over 15-30 minutes or SC on days 36-39 and 43-46; and thioguanine PO on days 36-49.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Nelarabine; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group I Arm II (Interim maintenance chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV and escalating doses of methotrexate IV on days 1, 11, 21, 31, and 41; pegaspargase* IM or IV over 1-2 hours on days 2 and 22; and methotrexate IT on days 1 and 31.
  Note: *Patients with an allergy to pegaspargase receive Erwinia asparaginase on Monday, Wednesday and Friday for two consecutive weeks starting the day of asparaginase substitution.
  Interventions: Drug: Asparaginase; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine Sulfate
- Group I Arm II (Maintenance chemotherapy) (Active Comparator): Patients receive vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, methotrexate IT, and nelarabine in Cycles 1, 2 and 3. Patients then receive treatment (without nelarabine) as follows: vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, and methotrexate IT as in arm II. Treatment (without nelarabine) repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 121) (for girls with T-ALL), and for those with T-LLY, and 3 years from the start of interim maintenance therapy (approximately week 173) (for boys with T-ALL).
  Interventions: Drug: Mercaptopurine; Drug: Methotrexate; Drug: Nelarabine; Drug: Prednisone; Drug: Vincristine Sulfate
- Group I Arm III (Consolidation chemotherapy) (Active Comparator): Patients receive methotrexate IT on days 1, 8, 15, and 22; cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine IV over 15-30 minutes or SC on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO on days 1-14 and 29-42; vincristine sulfate IV on days 15, 22, 43 and 50; and pegaspargase IM or IV over 1-2 hours on days 15 and 43. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 11-12, 15-19, and 22-26. (DS patients excluded as of 09/29/10.) Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT (1,200 cGy/dose) QD on days 15-21 and 22-28. Patients with low-risk disease do not undergo CRT.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Group I Arm III (Delayed intensification chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV on days 1, 8, 15, 43, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age and for patients with DS); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6, AND day 43; methotrexate IT on days 1, 29, and 36; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 15-30 minutes or SC on days 29-32 and 36-39; and thioguanine PO on days 29-42. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose (DS patients excluded as of 09/29/10).
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group I Arm III (Interim maintenance chemotherapy) (Active Comparator): Patients receive HDMTX IV over 24 hours and vincristine sulfate IV on days 1, 15, 29, and 43; mercaptopurine PO on days 1-56; and methotrexate IT on days 1 and 29. Beginning 42 hours after the start of HDMTX, patients also receive leucovorin calcium IV or PO once every 6 hours for 3 doses.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Vincristine Sulfate
- Group I Arm III (Maintenance chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV on days 1, 29, and 57; prednisone PO BID on days 1-5, 29-33, and 57-61; mercaptopurine PO QD on days 1-84; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; and methotrexate IT on day 1. Treatment repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 119) (for girls with T-ALL) and all patients with T-LLy, and 3 years from the start of interim maintenance therapy (approximately week 171) (for boys with T-ALL).
  Interventions: Drug: Methotrexate; Drug: Prednisone; Drug: Vincristine Sulfate
- Group I Arm IV (Delayed intensification chemotherapy) (Active Comparator): Patients receive vincristine sulfate IV on days 1, 8, 15, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age); doxorubicin IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6 AND day 50; methotrexate IT on days 1, 36, and 43; nelarabine IV over 60 minutes on days 29-33; cyclophosphamide IV over 30 minutes on day 36; cytarabine IV over 15-30 minutes or SC on days 36-39 and 43-46; and thioguanine PO on days 36-49.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Methotrexate; Drug: Nelarabine; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group I Arm IV (Interim maintenance chemotherapy) (Active Comparator): Patients receive HDMTX IV over 24 hours and vincristine IV on days 1, 15, 29, and 43; mercaptopurine PO on days 1-56; and methotrexate IT on days 1 and 29. Beginning 42 hours after the start of HDMTX, patients also receive leucovorin calcium IV or PO once every 6 hours for 3 doses.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Vincristine Sulfate
- Group I Arm IV (Maintenance chemotherapy) (Active Comparator): Patients receive vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, methotrexate IT, and nelarabine in Cycles 1, 2 and 3. Patients then receive treatment (without nelarabine) as follows: vincristine, prednisone, mercaptopurine, methotrexate PO, and methotrexate IT as in arm II. Treatment (without nelarabine) repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 121) (for girls with T-ALL), and for those with T-LLY, and 3 years from the start of interim maintenance therapy (approximately week 173) (for boys with T-ALL).
  Interventions: Drug: Mercaptopurine; Drug: Methotrexate; Drug: Nelarabine; Drug: Prednisone; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Asparaginase — Given IM or IV
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine Amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
  Arms: Group I Arm II (Interim maintenance chemotherapy)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Group 1 Arm IV (Consolidation chemotherapy); Group I Arm I (Consolidation chemotherapy); Group I Arm I (Delayed intensification chemotherapy; Group I Arm II (Consolidation chemotherapy); Group I Arm II (Delayed intensification chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm IV (Delayed intensification chemotherapy)
Drug: Cytarabine — Given IT, IV, or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Group 0 Induction Therapy; Group 1 Arm IV (Consolidation chemotherapy); Group I Arm I (Consolidation chemotherapy); Group I Arm I (Delayed intensification chemotherapy; Group I Arm II (Consolidation chemotherapy); Group I Arm II (Delayed intensification chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm IV (Delayed intensification chemotherapy)
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Group 0 Induction Therapy
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Group I Arm I (Delayed intensification chemotherapy; Group I Arm II (Delayed intensification chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm IV (Delayed intensification chemotherapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Group I Arm I (Delayed intensification chemotherapy; Group I Arm II (Delayed intensification chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm IV (Delayed intensification chemotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Group I Arm I (Maintenance chemotherapy); Group I Arm III (Interim maintenance chemotherapy); Group I Arm IV (Interim maintenance chemotherapy)
Drug: Leucovorin Calcium — Given PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Group I Arm I (Consolidation chemotherapy); Group I Arm I (Delayed intensification chemotherapy; Group I Arm I (Interim maintenance chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm III (Interim maintenance chemotherapy); Group I Arm IV (Interim maintenance chemotherapy)
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Group 1 Arm IV (Consolidation chemotherapy); Group I Arm I (Consolidation chemotherapy); Group I Arm I (Maintenance chemotherapy); Group I Arm II (Consolidation chemotherapy); Group I Arm II (Maintenance chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Interim maintenance chemotherapy); Group I Arm IV (Interim maintenance chemotherapy); Group I Arm IV (Maintenance chemotherapy)
Drug: Methotrexate — Given IT or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Group 0 Induction Therapy; Group 1 Arm IV (Consolidation chemotherapy); Group I Arm I (Consolidation chemotherapy); Group I Arm I (Delayed intensification chemotherapy; Group I Arm I (Interim maintenance chemotherapy); Group I Arm I (Maintenance chemotherapy); Group I Arm II (Consolidation chemotherapy); Group I Arm II (Interim maintenance chemotherapy); Group I Arm II (Maintenance chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm III (Interim maintenance chemotherapy); Group I Arm III (Maintenance chemotherapy); Group I Arm IV (Delayed intensification chemotherapy); Group I Arm IV (Interim maintenance chemotherapy); Group I Arm IV (Maintenance chemotherapy)
Drug: Nelarabine — Given IV
  Other Names: 2-Amino-6-methoxypurine arabinoside; 506U78; Arranon; Compound 506U78; GW506U78
  Arms: Group 1 Arm IV (Consolidation chemotherapy); Group I Arm II (Consolidation chemotherapy); Group I Arm II (Delayed intensification chemotherapy); Group I Arm II (Maintenance chemotherapy); Group I Arm IV (Delayed intensification chemotherapy); Group I Arm IV (Maintenance chemotherapy)
Drug: Pegaspargase — Given IM or IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
  Arms: Group 0 Induction Therapy; Group 1 Arm IV (Consolidation chemotherapy); Group I Arm I (Consolidation chemotherapy); Group I Arm I (Delayed intensification chemotherapy; Group I Arm I (Interim maintenance chemotherapy); Group I Arm II (Consolidation chemotherapy); Group I Arm II (Delayed intensification chemotherapy); Group I Arm II (Interim maintenance chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm IV (Delayed intensification chemotherapy)
Drug: Prednisone — Given IV or PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Group 0 Induction Therapy; Group I Arm I (Maintenance chemotherapy); Group I Arm II (Maintenance chemotherapy); Group I Arm III (Maintenance chemotherapy); Group I Arm IV (Maintenance chemotherapy)
Radiation: Radiation Therapy — Some patients undergo testicular and/or prophylactic cranial RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group 1 Arm IV (Consolidation chemotherapy); Group I Arm I (Consolidation chemotherapy); Group I Arm II (Consolidation chemotherapy); Group I Arm III (Consolidation chemotherapy)
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Group I Arm I (Delayed intensification chemotherapy; Group I Arm II (Delayed intensification chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm IV (Delayed intensification chemotherapy)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Group 0 Induction Therapy; Group I Arm I (Consolidation chemotherapy); Group I Arm I (Delayed intensification chemotherapy; Group I Arm I (Interim maintenance chemotherapy); Group I Arm I (Maintenance chemotherapy); Group I Arm II (Consolidation chemotherapy); Group I Arm II (Delayed intensification chemotherapy); Group I Arm II (Interim maintenance chemotherapy); Group I Arm II (Maintenance chemotherapy); Group I Arm III (Consolidation chemotherapy); Group I Arm III (Delayed intensification chemotherapy); Group I Arm III (Interim maintenance chemotherapy); Group I Arm III (Maintenance chemotherapy); Group I Arm IV (Delayed intensification chemotherapy); Group I Arm IV (Interim maintenance chemotherapy); Group I Arm IV (Maintenance chemotherapy)

SUMMARY:
This randomized phase III trial is studying different combination chemotherapy regimens and their side effects and comparing how well they work in treating young patients with newly diagnosed T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma. After a common induction therapy, patients were risk assigned and eligible for one or both post-induction randomizations: Escalating dose Methotrexate versus High Dose Methotrexate in Interim Maintenance therapy, No Nelarabine versus Nelarabine in Consolidation therapy. T-ALL patients are risk assigned as Low Risk, Intermediate Risk or High Risk. Low Risk patients are not eligible for the Nelarabine randomization, Patients with CNS disease at diagnosis were assgined to receive High Dose Methotrexate, patients who failed induction therapy were assigned to receive Nelarabine and High Dose Methotrexate. T-LLy patients were all assigned to escalating dose Methotrexate and were risk assigned as Standard Risk, High Risk and induction failures. Standard risk patients did not receive nelarabine, High risk T-LLy patients were randomized to No Nelarabine versus Nelarabine, and Induction failures were assigned to receive Nelarabine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine, through randomization, the relative safety and efficacy of the addition of nelarabine (Compound 506U78) to augmented Berlin-Frankfurt-Münster (BFM) therapy (Regimen C, Children's Cancer Group [CCG]-1961).

II. To determine the relative safety and efficacy of high dose methotrexate (5 g/m^2) with leucovorin (leucovorin calcium) rescue compared to escalating methotrexate without leucovorin rescue plus pegaspargase (Capizzi I) delivered during interim maintenance.

III. To gain preliminary data on the use of nelarabine in patients with high risk T-cell lymphoblastic lymphoma and its effect on long-term survival.

SECONDARY OBJECTIVES:

I. To determine the relative safety and efficacy of withholding radiation in patients with low risk T-cell acute lymphoblastic leukemia (T-ALL), while treating Intermediate and high risk patients with 1200 cGy of prophylactic cranial radiation.

OUTLINE: This is a randomized, controlled, factorial-group, multicenter study.

GROUP 0 (INDUCTION THERAPY): All patients (T-ALL and T-LLy) receive cytarabine intrathecally (IT) on day 1; vincristine sulfate intravenously (IV) on days 1, 8, 15, and 22; prednisone IV or orally (PO) twice daily (BID) on days 1-28; pegaspargase intramuscularly (IM) (may give IV over 1 to 2 hours) on day 4, 5, or 6; duanorubicin IV on days 1, 8, 15 and 22; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease).

GROUP I ARM I COMBINATION CHEMOTHERAPY (CONSOLIDATION CHEMOTHERAPY): Patients receive methotrexate IT on days 1, 8, 15, and 22; cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine IV over 15-30 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO on days 1-14 and 29-42; vincristine sulfate IV on days 15, 22, 43 and 50; and pegaspargase IM or IV over 1-2 hours on days 15 and 43. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 11-12, 15-19, and 22-26. (DS patients excluded as of 09/29/10.) Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT (1,200 cGy/dose) QD on days 15-21 and 22-28. Patients with low-risk disease do not undergo conformal radiation therapy (CRT). Patients with standard risk T-LLy received Arm I, and those with high risk T-LLy were randomized between Arm I and Arm II combination chemotherapy.

GROUP I ARM I COMBINATION CHEMOTHERAPY (DELAYED INTENSIFICATION CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 8, 15, 43, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age and for patients with DS); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6, AND day 43; methotrexate IT on days 1, 29, and 36; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 15-30 minutes or SC on days 29-32 and 36-39; and thioguanine PO on days 29-42. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose (DS patients excluded as of 09/29/10). Standard risk T-LLy patients were assigned to Arm I and those with high risk were randomized between Arm I and Arm II.

GROUP I ARM I COMBINATION CHEMOTHERAPY (INTERIM MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate IV and escalating doses of methotrexate IV on days 1, 11, 21, 31, and 41; pegaspargase* IM or IV over 1-2 hours on days 2 and 22; and methotrexate IT on days 1 and 31. Patients with DS also receive leucovorin calcium PO 48 and 60 hours after each methotrexate IT dose (DS patients excluded as of 09/29/10).

Note: *Patients with an allergy to pegaspargase receive Erwinia asparaginase on days 2, 4, 6, 8, 10, 12, 22, 24, 26, 28, 30, and 32.

GROUP I ARM I COMBINATION CHEMOTHERAPY (MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 29, and 57; prednisone PO BID on days 1-5, 29-33, and 57-61; mercaptopurine PO QD on days 1-84; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; and methotrexate IT on day 1. Treatment repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 119) (for girls with T-ALL), all patients with T-LLy, and 3 years from the start of interim maintenance therapy (approximately week 171) (for boys with T-ALL).

GROUP I ARM II COMBINATION CHEMOTHERAPY (CONSOLIDATION CHEMOTHERAPY): Patients receive nelarabine IV over 60 minutes on days 1-5 and 43-47; methotrexate IT on days 15, 22, 57, and 64; cyclophosphamide IV over 30 minutes on days 8 and 50; cytarabine IV over 15-30 minutes or SC on days 8-11, 15-18, 50-53 and 57-60; mercaptopurine PO on days 8-21 and 50-63; vincristine sulfate IV on days 22, 29, 64, and 71; and pegaspargase IM or IV over 1-2 hours on days 22 and 64. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 15, 22-26, and 29-33 (DS patients excluded as of 09/29/10). (Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT QD on days 22-28 and 29-35. Patients with high risk T-LLy were either randomized to Arm I or Arm II. Patients with T-LLy who failed induction therapy were assigned to Arm II.

GROUP I ARM II COMBINATION CHEMOTHERAPY (DELAYED INTENSIFICATION CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 8, 15, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6 AND day 50; methotrexate IT on days 1, 36, and 43; nelarabine IV over 60 minutes on days 29-33; cyclophosphamide IV over 30 minutes on day 36; cytarabine IV over 15-30 minutes or SC on days 36-39 and 43-46; and thioguanine PO on days 36-49.

GROUP I ARM II COMBINATION CHEMOTHERAPY (INTERIM MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate IV and escalating doses of methotrexate IV on days 1, 11, 21, 31, and 41; pegaspargase* IM or IV over 1-2 hours on days 2 and 22; and methotrexate IT on days 1 and 31.

Note: *Patients with an allergy to pegaspargase receive Erwinia asparaginase on Monday, Wednesday and Friday for two consecutive weeks starting the day of asparaginase substitution.

GROUP I ARM II COMBINATION CHEMOTHERAPY (MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, methotrexate IT, and nelarabine in Cycles 1, 2 and 3. Patients then receive treatment (without nelarabine) as follows: vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, and methotrexate IT as in arm II. Treatment (without nelarabine) repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 121) (for girls with T-ALL), and for those with T-LLY, and 3 years from the start of interim maintenance therapy (approximately week 173) (for boys with T-ALL).

GROUP I ARM III COMBINATION CHEMOTHERAPY (CONSOLIDATION CHEMOTHERAPY): Patients receive methotrexate IT on days 1, 8, 15, and 22; cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine IV over 15-30 minutes or SC on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO on days 1-14 and 29-42; vincristine sulfate IV on days 15, 22, 43 and 50; and pegaspargase IM or IV over 1-2 hours on days 15 and 43. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose. Patients with persistent testicular disease or with DS and testicular disease undergo testicular radiotherapy on days 11-12, 15-19, and 22-26. (DS patients excluded as of 09/29/10.) Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT (1,200 cGy/dose) QD on days 15-21 and 22-28. Patients with low-risk disease do not undergo CRT.

GROUP I ARM III COMBINATION CHEMOTHERAPY (DELAYED INTENSIFICATION CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 8, 15, 43, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age and for patients with DS); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6, AND day 43; methotrexate IT on days 1, 29, and 36; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 15-30 minutes or SC on days 29-32 and 36-39; and thioguanine PO on days 29-42. Patients with DS also receive leucovorin calcium PO at 48 and 60 hours after each methotrexate dose (DS patients excluded as of 09/29/10).

GROUP I ARM III COMBINATION CHEMOTHERAPY (INTERIM MAINTENANCE CHEMOTHERAPY): Patients receive high dose methotrexate (HDMTX) IV over 24 hours and vincristine sulfate IV on days 1, 15, 29, and 43; mercaptopurine PO on days 1-56; and methotrexate IT on days 1 and 29. Beginning 42 hours after the start of HDMTX, patients also receive leucovorin calcium IV or PO once every 6 hours for 3 doses.

GROUP I ARM III COMBINATION CHEMOTHERAPY (MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 29, and 57; prednisone PO BID on days 1-5, 29-33, and 57-61; mercaptopurine PO QD on days 1-84; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; and methotrexate IT on day 1. Treatment repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 119) (for girls with T-ALL) and all patients with T-LLy, and 3 years from the start of interim maintenance therapy (approximately week 171) (for boys with T-ALL).

GROUP I ARM IV COMBINATION CHEMOTHERAPY (CONSOLIDATION CHEMOTHERAPY): Patients receive nelarabine IV over 60 minutes on days 1-5 and 43-47; methotrexate IT on days 15, 22, 57, and 64; cyclophosphamide IV over 30 minutes on days 8 and 50; cytarabine IV over 15-30 minutes or SC on days 8-11, 15-18, 50-53 and 57-60; mercaptopurine PO on days 8-21 and 50-63; vincristine sulfate IV on days 22, 29, 64, and 71; and pegaspargase IM or IV over 1-2 hours on days 22 and 64. (DS patients excluded as of 09/29/10). (Patients with intermediate-risk or high-risk disease (CNS1 or CNS2) undergo prophylactic CRT QD on days 22-28 and 29-35.

GROUP I ARM IV COMBINATION CHEMOTHERAPY (DELAYED INTENSIFICATION CHEMOTHERAPY): Patients receive vincristine sulfate IV on days 1, 8, 15, and 50; dexamethasone IV or PO BID on days 1-21 (for patients < 10 years of age) OR on days 1-7 and 15-21 (for patients >= 10 years of age); doxorubicin hydrochloride IV on days 1, 8, and 15; pegaspargase IM or IV over 1-2 hours on day 4, 5, OR 6 AND day 50; methotrexate IT on days 1, 36, and 43; nelarabine IV over 60 minutes on days 29-33; cyclophosphamide IV over 30 minutes on day 36; cytarabine IV over 15-30 minutes or SC on days 36-39 and 43-46; and thioguanine PO on days 36-49.

GROUP I ARM IV COMBINATION CHEMOTHERAPY (INTERIM MAINTENANCE CHEMOTHERAPY): Patients receive HDMTX IV over 24 hours and vincristine sulfate IV on days 1, 15, 29, and 43; mercaptopurine PO on days 1-56; and methotrexate IT on days 1 and 29. Beginning 42 hours after the start of HDMTX, patients also receive leucovorin calcium IV or PO once every 6 hours for 3 doses.

GROUP I ARM IV COMBINATION CHEMOTHERAPY (MAINTENANCE CHEMOTHERAPY): Patients receive vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, methotrexate IT, and nelarabine in Cycles 1, 2 and 3. Patients then receive treatment (without nelarabine) as follows: vincristine sulfate, prednisone, mercaptopurine, methotrexate PO, and methotrexate IT as in arm II. Treatment (without nelarabine) repeats every 84 days until the total duration of study treatment is 2 years from the start of interim maintenance therapy (approximately week 121) (for girls with T-ALL), and for those with T-LLY, and 3 years from the start of interim maintenance therapy (approximately week 173) (for boys with T-ALL).

After completion of study therapy, patients are followed periodically for at least 10 years.

ELIGIBILITY:
Inclusion Criteria:

* T-ALL patients must be enrolled on AALL08B1 prior to treatment and enrollment on AALL0434
* Patients must have newly diagnosed T-ALL or T-lineage lymphoblastic lymphoma (T-NHL) stage II-IV; B-lineage lymphoblastic lymphoma will not be eligible for this study; a diagnosis of T-ALL is established when leukemic blasts lack myeloperoxidase or evidence of B-lineage derivation (cluster of differentiation [CD]19/CD22/CD20), and express either surface or cytoplasmic CD3 or two or more of the antigens CD8, CD7, CD5, CD4, CD2 or CD1a; if surface CD3 is expressed on all leukemic cells, additional markers of immaturity, including transmission disequilibrium test (TdT), CD34 or CD99 will be assessed for expression; cases with uncertain expression will receive additional review within the appropriate Children's Oncology Group (COG) reference laboratory
* T-NHL PATIENTS:

  * For T-NHL patients with tissue available for flow cytometry, the criterion for diagnosis should be analogous to T-ALL; for tissue processed by other means (i.e. paraffin blocks), the methodology and criteria for immunophenotypic analysis to establish the diagnosis of T-NHL defined by the submitting institution will be accepted
* Prior therapy restrictions

  * Patients shall have had no prior cytotoxic chemotherapy with the exception of steroids and/or IT cytarabine
  * IT chemotherapy with cytarabine is allowed prior to registration for patient convenience; this is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture; (Note: the CNS status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment); systemic chemotherapy must begin within 72 hours of this IT therapy
  * Patients diagnosed as having T-NHL or T-ALL with respiratory distress or hyperleukocytosis may require steroids prior to the initiation of additional systemic therapy; they are eligible for AALL0434 and will be stratified, based on the initial complete blood count (CBC); steroid pretreatment may alter the risk group assessment; if the T-ALL patient's clinical status precludes a lumbar puncture within 48 hours of the initiation of steroid therapy, T-ALL patients CANNOT be classified as low risk and will be Intermediate or high risk based on the results of the day 29 marrow as above; patients with T-NHL who receive steroid pre-treatment will be classified as high risk; the dose and duration of previous steroid therapy should be carefully documented
  * For the management of airway compromise, patients who have received emergent chest irradiation up to 600 cGy will be eligible for this study
* Patients with a prior seizure disorder requiring anti-convulsant therapy are not eligible to receive nelarabine; in addition, patients with pre-existing grade 2 (or greater) peripheral neurotoxicity, as determined prior to Induction treatment by the treating physician or a neurologist, are not eligible to receive nelarabine; these restrictions in eligibility are designed to prevent excessive nelarabine-induced central and peripheral neurotoxicity in at-risk patients; for the purposes of this study, this includes any patient that has received anticonvulsant therapy to prevent/treat seizures in the prior two years

Exclusion Criteria:

* Pregnant or lactating females are ineligible
* Patients with Down syndrome are ineligible to enroll onto this study
* For T-NHL patients the following additional exclusion criteria apply:

  * B-precursor lymphoblastic lymphoma
  * Morphologically unclassifiable lymphoma
  * Absence of both B-cell and T-cell phenotype markers in a case submitted as lymphoblastic lymphoma
  * CNS3-positive or testicular involvement

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1895 (Actual)
Dates: Start 2007-01-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart S Winter, Principal Investigator — Children's Oncology Group
Locations (215):
- United States (191):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Switzerland (2):
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Derived] Wood BL, Devidas M, Summers RJ, Chen Z, Asselin B, Rabin KR, Zweidler-McKay PA, Winick NJ, Borowitz MJ, Carroll WL, Raetz EA, Loh ML, Hunger SP, Dunsmore KP, Teachey DT, Winter SS. Prognostic significance of ETP phenotype and minimal residual disease in T-ALL: a Children's Oncology Group study. Blood. 2023 Dec 14;142(24):2069-2078. doi: 10.1182/blood.2023020678. PMID 37556734
- [Derived] Gossai NP, Devidas M, Chen Z, Wood BL, Zweidler-McKay PA, Rabin KR, Loh ML, Raetz EA, Winick NJ, Burke MJ, Carroll AJ, Esiashvili N, Heerema NA, Carroll WL, Hunger SP, Dunsmore KP, Winter SS, Teachey DT. Central nervous system status is prognostic in T-cell acute lymphoblastic leukemia: a Children's Oncology Group report. Blood. 2023 Apr 13;141(15):1802-1811. doi: 10.1182/blood.2022018653. PMID 36603187
- [Derived] Gaynon PS, Parekh C. A new standard of care for childhood T-cell acute lymphoblastic leukemia? Pediatr Blood Cancer. 2021 Oct;68(10):e29238. doi: 10.1002/pbc.29238. Epub 2021 Jul 24. No abstract available. PMID 34302711
- [Derived] Dunsmore KP, Winter SS, Devidas M, Wood BL, Esiashvili N, Chen Z, Eisenberg N, Briegel N, Hayashi RJ, Gastier-Foster JM, Carroll AJ, Heerema NA, Asselin BL, Rabin KR, Zweidler-Mckay PA, Raetz EA, Loh ML, Schultz KR, Winick NJ, Carroll WL, Hunger SP. Children's Oncology Group AALL0434: A Phase III Randomized Clinical Trial Testing Nelarabine in Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia. J Clin Oncol. 2020 Oct 1;38(28):3282-3293. doi: 10.1200/JCO.20.00256. Epub 2020 Aug 19. PMID 32813610
- [Derived] Hayashi RJ, Winter SS, Dunsmore KP, Devidas M, Chen Z, Wood BL, Hermiston ML, Teachey DT, Perkins SL, Miles RR, Raetz EA, Loh ML, Winick NJ, Carroll WL, Hunger SP, Lim MS, Gross TG, Bollard CM. Successful Outcomes of Newly Diagnosed T Lymphoblastic Lymphoma: Results From Children's Oncology Group AALL0434. J Clin Oncol. 2020 Sep 10;38(26):3062-3070. doi: 10.1200/JCO.20.00531. Epub 2020 Jun 17. PMID 32552472
- [Derived] Winter SS, Dunsmore KP, Devidas M, Wood BL, Esiashvili N, Chen Z, Eisenberg N, Briegel N, Hayashi RJ, Gastier-Foster JM, Carroll AJ, Heerema NA, Asselin BL, Gaynon PS, Borowitz MJ, Loh ML, Rabin KR, Raetz EA, Zweidler-Mckay PA, Winick NJ, Carroll WL, Hunger SP. Improved Survival for Children and Young Adults With T-Lineage Acute Lymphoblastic Leukemia: Results From the Children's Oncology Group AALL0434 Methotrexate Randomization. J Clin Oncol. 2018 Oct 10;36(29):2926-2934. doi: 10.1200/JCO.2018.77.7250. Epub 2018 Aug 23. PMID 30138085
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were stratified between the 2 disease groups (T-ALL and T-LLy) for Induction and then risk assigned treatment based upon the patient's response.
Groups:
- T-ALL Induction Therapy: All patients diagnosed as T-ALL for induction
- T-LLy Induction Therapy: All patients diagnosed as T-LLy for induction
- T-ALL: Capizzi MTX Without Nelarabine: T-All patients who received Capizzi MTX without Nelarabine
- T-ALL: Capizzi MTX With Nelarabine: T-All patients who received Capizzi MTX with Nelarabine
- T-ALL: High Dose MTX Without Nelarabine: T-All patients who received High Dose MTX without Nelarabine
- T-ALL: High Dose MTX With Nelarabine: T-All patients who received High Dose MTX with Nelarabine
- T-LLy: Capizzi MTX Without Nelarabine: T-LLy patients who received Capizzi MTX without Nelarabine
- T-LLy: Capizzi MTX With Nelarabine: T-LLy patients who received Capizzi MTX with Nelarabine
Period: Induction
Arm/Group | T-ALL Induction Therapy | T-LLy Induction Therapy | T-ALL: Capizzi MTX Without Nelarabine | T-ALL: Capizzi MTX With Nelarabine | T-ALL: High Dose MTX Without Nelarabine | T-ALL: High Dose MTX With Nelarabine | T-LLy: Capizzi MTX Without Nelarabine | T-LLy: Capizzi MTX With Nelarabine
Started | 1596 | 299 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1189 | 205 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 407 | 94 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 19 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 83 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 33 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal of Further Protocol Therapy | 225 | 44 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Entered another COG therapeutic protocol | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient transferred Tx to Non-COG Site | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Identified as Philadelphia Chr. Positive | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inevaluable | 18 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to Complete Randomization | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Hematopoietic Stem Cell Transplantation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Recurrent leukemia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post Induction Therapy by Tx Assignment
Arm/Group | T-ALL Induction Therapy | T-LLy Induction Therapy | T-ALL: Capizzi MTX Without Nelarabine | T-ALL: Capizzi MTX With Nelarabine | T-ALL: High Dose MTX Without Nelarabine | T-ALL: High Dose MTX With Nelarabine | T-LLy: Capizzi MTX Without Nelarabine | T-LLy: Capizzi MTX With Nelarabine
Started | 0 | 0 | 372 | 147 | 451 | 219 | 143 | 62
Low Risk | 0 | 0 | 217 | 0 | 55 | 0 | 0 | 0
Intermediate Risk | 0 | 0 | 99 | 95 | 257 | 93 | 0 | 0
High Risk | 0 | 0 | 56 | 52 | 55 | 52 | 0 | 0
CNS 3 and/or Testicular Disease | 0 | 0 | 0 | 0 | 84 | 31 | 0 | 0
T-ALL M3 Marrow End of Induction | 0 | 0 | 0 | 0 | 0 | 43 | 0 | 0
T-LLy Standard Risk | 0 | 0 | 0 | 0 | 0 | 0 | 82 | 0
T-LLy High Risk | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 60
T-LLy Induction Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Completed | 0 | 0 | 287 | 103 | 319 | 118 | 115 | 48
Not Completed | 0 | 0 | 85 | 44 | 132 | 101 | 28 | 14
Not completed — Adverse Event | 0 | 0 | 7 | 4 | 8 | 12 | 2 | 0
Not completed — Death | 0 | 0 | 3 | 0 | 5 | 5 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 24 | 19 | 27 | 45 | 10 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Refusal of Further Protocol Therapy | 0 | 0 | 27 | 10 | 36 | 16 | 4 | 2
Not completed — Entered another COG therapeutic protocol | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Patient transferred Tx to Non-COG Site | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 7
Not completed — Inevaluable | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0
Not completed — Hematopoietic Stem Cell Transplantation | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Recurrent Leukemia After Total Remission | 0 | 0 | 13 | 7 | 49 | 15 | 1 | 0
Not completed — Development of SMN | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T-ALL Induction Therapy | T-LLy Induction Therapy | Total
Number analyzed (Participants) | 1596 | 299 | 1895
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1493 | 268 | 1761
  Between 18 and 65 years | 103 | 31 | 134
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.05 (5.3) | 11.13 (5.8) | 10.22 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 407 | 90 | 497
  Male | 1189 | 209 | 1398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 227 | 45 | 272
  Not Hispanic or Latino | 1307 | 244 | 1551
  Unknown or Not Reported | 62 | 10 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 1 | 7
  Asian | 87 | 11 | 98
  Native Hawaiian or Other Pacific Islander | 12 | 4 | 16
  Black or African American | 204 | 50 | 254
  White | 1122 | 208 | 1330
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 165 | 25 | 190

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) for Randomized Nelarabine T-ALL Cohort (Arm I vs. Arm II vs. Arm III vs. Arm IV)
Description: Disease Free Probability where DFS time is defined as time from randomization end of induction to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free.
Time Frame: 4 years from randomization at the end of induction
Population: Includes only T-cell Acute Lymphoblastic Leukemia (T-ALL) patients randomized to Nelarabine versus No Nelarabine. T-LLY patients are excluded from this analysis. Induction failures non-randomly assigned to Arm IV were excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- ARM I (Combination Chemotherapy): No Nelarabine, Capizzi Methotrexate
- ARM II (Combination Chemotherapy): Nelarabine, Capizzi Methotrexate
- ARM III (Combination Chemotherapy): No Nelarabine, High-Dose Methotrexate
- ARM IV (Combination Chemotherapy): Nelarabine, High-Dose Methotrexate
Arm/Group | ARM I (Combination Chemotherapy) | ARM II (Combination Chemotherapy) | ARM III (Combination Chemotherapy) | ARM IV (Combination Chemotherapy)
Number analyzed (Participants) | 151 | 147 | 185 | 176
percent probability | 89.01 [83.4 to 94.6] | 90.53 [85.0 to 96.0] | 78.07 [71.2 to 84.9] | 86.46 [80.6 to 92.4]

2. Primary Outcome: Disease-free Survival (DFS) for Randomized Nelarabine T-ALL Cohort (Arm I + Arm III vs. Arm II + Arm IV)
Description: Disease Free Probability where DFS time is defined as time from randomization end of induction to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event
Time Frame: 4 years from randomization at the end of induction
Population: Includes subjects randomized to Nelarabine versus No Nelarabine
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- ARM I and ARM III (Combination Chemotherapy): No Nelarabine (Combined)
- ARM II and ARM IV (Combination Chemotherapy): Nelarabine (Combined)
Arm/Group | ARM I and ARM III (Combination Chemotherapy) | ARM II and ARM IV (Combination Chemotherapy)
Number analyzed (Participants) | 336 | 323
percent probability | 82.96 [78.4 to 87.5] | 88.30 [84.2 to 92.4]

3. Primary Outcome: Disease-free Survival (DFS) for Randomized Methotrexate T-ALL Cohort (Arm I vs. Arm II vs. Arm III vs. Arm IV)
Description: Disease-free survival defined as time from randomization end of induction to first event (relapse, second malignant neoplasm, remission death) or date of last contact for those who are event-free.
Time Frame: 4 years from randomization at the end of induction
Population: Includes only T-cell Acute Lymphoblastic Leukemia (T-ALL) patients randomized to Capizzi Methotrexate (CMTX) versus High-Dose Methotrexate (HDMTX). CNS3 patients non-randomly assigned to HDMTX (Arms III and IV) and Induction failures non-randomly assigned to Arm IV were excluded. T-LLY patients are excluded.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | ARM I (Combination Chemotherapy) | ARM II (Combination Chemotherapy) | ARM III (Combination Chemotherapy) | ARM IV (Combination Chemotherapy)
Number analyzed (Participants) | 372 | 147 | 367 | 145
percent probability | 91.76 [88.8 to 94.8] | 90.53 [85.0 to 96.0] | 86.06 [82.2 to 89.9] | 84.89 [78.0 to 91.8]

4. Primary Outcome: Disease-free Survival (DFS) for Randomized Methotrexate T-ALL Cohort (Arm I + Arm II vs. Arm III + Arm IV)
Description: as for outcome 1
Time Frame: 4 years from randomization at the end of induction
Population: Includes subjects randomized to Capizzi Methotrexate versus High-Dose Methotrexate
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- ARM I and ARM II (Combination Chemotherapy): Capizzi Methotrexate (Combined)
- ARM III and ARM IV (Combination Chemotherapy): High-Dose Methotrexate (Combined)
Arm/Group | ARM I and ARM II (Combination Chemotherapy) | ARM III and ARM IV (Combination Chemotherapy)
Number analyzed (Participants) | 519 | 512
percent probability | 91.45 [88.8 to 94.1] | 85.78 [82.4 to 89.1]

5. Primary Outcome: Disease-free Survival (DFS) for T-cell Lymphoblastic Lymphoma (T-LLy) Cohort
Description: as for outcome 1
Time Frame: 4 years from end of induction
Population: Includes T-cell lymphoblastic lymphoma (T-LLy) patients that are standard risk, high risk and induction failures. All Standard risk T-LLy patients only received Arm I. Induction failures were assigned to Arm II.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | ARM I (Combination Chemotherapy) | ARM II (Combination Chemotherapy)
Number analyzed (Participants) | 143 | 62
percent probability
  Standard Risk: number analyzed (Participants) | 82 | 0
  Standard Risk | 87.4 [79.6 to 95.2] |
  High Risk: number analyzed (Participants) | 61 | 60
  High Risk | 85.1 [75.7 to 94.5] | 85.0 [75.0 to 95.0]
  Induction Failure: number analyzed (Participants) | 0 | 2
  Induction Failure |  | 100 [100 to 100]

6. Secondary Outcome: Cumulative Incidence of CNS Relapse for T-ALL by Risk Group
Description: Cumulative incidence of CNS relapse adjusting for DFS events, was calculated using the method Gray et. al. High risk patients receive cranial radiation and low risk patients receive no cranial radiation.
Time Frame: 4 years from randomization at the end of induction
Population: Includes only low risk, intermediate risk and high risk T-cell Acute Lymphoblastic Leukemia (T-ALL) subjects. There were no low risk participants on Arm II and Arm IV. Patients with CNS3, and Induction Failures are excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | ARM I (Combination Chemotherapy) | ARM II (Combination Chemotherapy) | ARM III (Combination Chemotherapy) | ARM IV (Combination Chemotherapy)
Number analyzed (Participants) | 372 | 147 | 451 | 176
percent probability
  Low Risk: number analyzed (Participants) | 54 | 0 | 55 | 0
  Low Risk | 1.85 [0 to 5.5] |  | 1.92 [0 to 5.7] |
  Intermediate Risk: number analyzed (Participants) | 262 | 95 | 333 | 118
  Intermediate Risk | 1.16 [0 to 2.5] | 1.08 [0 to 3.2] | 9.1 [6.0 to 12.2] | 0.85 [0 to 2.5]
  High Risk: number analyzed (Participants) | 56 | 52 | 63 | 58
  High Risk | 3.64 [0 to 8.6] | 0 [0 to 0] | 6.52 [0.3 to 12.8] | 3.45 [0 to 8.2]

ADVERSE EVENTS:
Time Frame: From start of Induction therapy to end of Maintenance therapy, up to 10 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Groups:
- T-ALL Post Induction Therapy: T-ALL patients who went off therapy at the end of induction, excluding patients who died at induction
- T-LLy Post Induction Therapy: T-LLy patients who went off therapy at the end of induction, excluding patients who died at induction
Arm/Group | T-ALL Induction Therapy | T-ALL Post Induction Therapy | T-ALL: Capizzi MTX Without Nelarabine | T-ALL: Capizzi MTX With Nelarabine | T-ALL: High Dose MTX Without Nelarabine | T-ALL: High Dose MTX With Nelarabine | T-LLy Induction Therapy | T-LLy Post Induction Therapy | T-LLy: Capizzi MTX Without Nelarabine | T-LLy: Capizzi MTX With Nelarabine
All-Cause Mortality (participants affected / at risk) | 6/1563 | 39/368 | 26/372 | 10/147 | 45/451 | 35/219 | 0/285 | 8/80 | 17/143 | 5/62
Serious Adverse Events (participants affected / at risk) | 25/1563 | 1/368 | 18/372 | 44/147 | 23/451 | 66/219 | 1/285 | 0/80 | 10/143 | 20/62
Other Adverse Events (participants affected / at risk) | 983/1563 | 0/368 | 357/372 | 134/147 | 436/451 | 197/219 | 152/285 | 4/80 | 140/143 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-ALL Induction Therapy (N=1563) | T-ALL Post Induction Therapy (N=368) | T-ALL: Capizzi MTX Without Nelarabine (N=372) | T-ALL: Capizzi MTX With Nelarabine (N=147) | T-ALL: High Dose MTX Without Nelarabine (N=451) | T-ALL: High Dose MTX With Nelarabine (N=219) | T-LLy Induction Therapy (N=285) | T-LLy Post Induction Therapy (N=80) | T-LLy: Capizzi MTX Without Nelarabine (N=143) | T-LLy: Capizzi MTX With Nelarabine (N=62)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 6 (8) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arachnoiditis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 6 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-ALL Induction Therapy (N=1563) | T-ALL Post Induction Therapy (N=368) | T-ALL: Capizzi MTX Without Nelarabine (N=372) | T-ALL: Capizzi MTX With Nelarabine (N=147) | T-ALL: High Dose MTX Without Nelarabine (N=451) | T-ALL: High Dose MTX With Nelarabine (N=219) | T-LLy Induction Therapy (N=285) | T-LLy Post Induction Therapy (N=80) | T-LLy: Capizzi MTX Without Nelarabine (N=143) | T-LLy: Capizzi MTX With Nelarabine (N=62)
Anemia (Blood and lymphatic system disorders) | 57 (60) | 0 (0) | 87 (139) | 26 (37) | 93 (142) | 25 (29) | 2 (2) | 0 (0) | 23 (33) | 9 (12)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 96 (101) | 0 (0) | 233 (504) | 87 (153) | 283 (614) | 102 (168) | 3 (3) | 2 (2) | 91 (160) | 27 (52)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asystole (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 22 (22) | 0 (0) | 28 (34) | 8 (13) | 19 (30) | 13 (15) | 3 (3) | 0 (0) | 6 (7) | 4 (6)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 0 (0) | 4 (4) | 2 (2) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 1 (3)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (18) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 0 (0) | 20 (21) | 7 (7) | 26 (27) | 8 (8) | 2 (2) | 0 (0) | 2 (2) | 2 (6)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 17 (17) | 0 (0) | 54 (64) | 19 (21) | 77 (83) | 35 (37) | 3 (3) | 0 (0) | 24 (28) | 9 (10)
Nausea (Gastrointestinal disorders) | 9 (9) | 0 (0) | 32 (37) | 14 (18) | 20 (25) | 17 (18) | 5 (5) | 0 (0) | 13 (15) | 6 (9)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 10 (12) | 1 (1) | 9 (9) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 0 (0) | 9 (9) | 10 (13) | 15 (19) | 8 (8) | 1 (1) | 2 (2) | 9 (9) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 12 (13) | 3 (3) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (14) | 0 (0) | 40 (51) | 14 (18) | 38 (47) | 19 (23) | 3 (3) | 0 (0) | 14 (16) | 9 (14)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 9 (10) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Fever (General disorders) | 12 (12) | 0 (0) | 49 (62) | 16 (18) | 42 (48) | 15 (17) | 1 (1) | 1 (1) | 10 (11) | 7 (9)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 9 (9) | 0 (0) | 5 (7) | 0 (0) | 10 (10) | 3 (3) | 4 (4) | 0 (0) | 6 (6) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 9 (9) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 3 (3) | 0 (0) | 17 (18) | 6 (6) | 18 (18) | 8 (9) | 0 (0) | 1 (1) | 10 (10) | 5 (5)
Anaphylaxis (Immune system disorders) | 3 (3) | 0 (0) | 40 (42) | 10 (10) | 51 (53) | 13 (13) | 0 (0) | 0 (0) | 10 (10) | 2 (2)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 6 (9) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 12 (13) | 0 (0) | 13 (17) | 3 (3) | 20 (27) | 9 (13) | 4 (4) | 0 (0) | 10 (12) | 3 (3)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 4 (4) | 0 (0) | 18 (19) | 2 (2) | 15 (17) | 7 (8) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 102 (127) | 0 (0) | 145 (280) | 41 (61) | 184 (298) | 53 (77) | 15 (17) | 0 (0) | 31 (35) | 8 (10)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 13 (14) | 0 (0) | 38 (44) | 12 (15) | 41 (52) | 14 (16) | 1 (1) | 0 (0) | 9 (9) | 4 (4)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 8 (8) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 9 (11) | 4 (4) | 19 (21) | 6 (6) | 0 (0) | 0 (0) | 8 (9) | 2 (2)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 13 (13) | 0 (0) | 7 (7) | 4 (5) | 7 (8) | 2 (3) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 15 (20) | 7 (7) | 16 (17) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 18 (19) | 0 (0) | 28 (33) | 8 (11) | 29 (29) | 13 (15) | 1 (1) | 0 (0) | 7 (8) | 3 (3)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (2) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Splenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 7 (8) | 0 (0) | 49 (63) | 17 (18) | 45 (55) | 20 (23) | 1 (1) | 0 (0) | 17 (23) | 8 (11)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 0 (0) | 15 (15) | 2 (2) | 10 (11) | 9 (11) | 1 (1) | 0 (0) | 8 (9) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 5 (6) | 0 (0) | 3 (4) | 0 (0) | 6 (7) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury to superior vena cava (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 12 (12) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 16 (16) | 0 (0) | 6 (8) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 133 (133) | 0 (0) | 157 (456) | 62 (166) | 182 (493) | 83 (217) | 25 (25) | 1 (1) | 49 (97) | 21 (50)
Alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0) | 7 (7) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 72 (72) | 0 (0) | 86 (133) | 35 (59) | 99 (145) | 36 (54) | 6 (6) | 1 (2) | 27 (40) | 10 (12)
Blood antidiuretic hormone abnormal (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 29 (29) | 0 (0) | 42 (66) | 20 (31) | 52 (85) | 20 (40) | 4 (4) | 1 (1) | 25 (29) | 6 (8)
Blood gonadotrophin abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood prolactin abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 4 (4) | 0 (0) | 3 (5) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 21 (21) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Fibrinogen decreased (Investigations) | 75 (76) | 0 (0) | 2 (2) | 3 (4) | 3 (5) | 1 (1) | 8 (8) | 1 (1) | 5 (5) | 0 (0)
GGT increased (Investigations) | 22 (22) | 0 (0) | 14 (27) | 3 (4) | 12 (24) | 6 (9) | 1 (1) | 0 (0) | 6 (8) | 1 (2)
Growth hormone abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 15 (15) | 0 (0) | 15 (19) | 9 (13) | 26 (31) | 4 (4) | 3 (3) | 1 (1) | 10 (12) | 3 (3)
Lymphocyte count decreased (Investigations) | 6 (6) | 0 (0) | 24 (41) | 9 (15) | 28 (44) | 13 (18) | 3 (3) | 0 (0) | 7 (13) | 3 (5)
Neutrophil count decreased (Investigations) | 97 (98) | 0 (0) | 276 (710) | 89 (189) | 331 (1010) | 116 (277) | 8 (8) | 1 (1) | 100 (208) | 35 (76)
Platelet count decreased (Investigations) | 61 (61) | 0 (0) | 117 (201) | 29 (44) | 150 (251) | 50 (75) | 1 (1) | 0 (0) | 37 (53) | 13 (19)
Serum amylase increased (Investigations) | 11 (11) | 0 (0) | 11 (13) | 2 (4) | 17 (17) | 5 (5) | 1 (1) | 1 (1) | 5 (5) | 1 (2)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 3 (3) | 0 (0) | 1 (6) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 17 (17) | 0 (0) | 23 (25) | 6 (6) | 16 (17) | 5 (5) | 5 (5) | 0 (0) | 6 (8) | 3 (3)
White blood cell decreased (Investigations) | 54 (54) | 0 (0) | 110 (253) | 35 (62) | 125 (353) | 40 (70) | 2 (2) | 0 (0) | 38 (61) | 11 (18)
Acidosis (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 27 (27) | 0 (0) | 38 (45) | 17 (35) | 32 (45) | 16 (21) | 4 (4) | 0 (0) | 12 (13) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 15 (15) | 0 (0) | 51 (62) | 22 (25) | 30 (34) | 15 (18) | 9 (9) | 0 (0) | 11 (13) | 7 (7)
Glucose intolerance (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 216 (217) | 0 (0) | 14 (16) | 4 (7) | 42 (67) | 14 (22) | 17 (18) | 0 (0) | 15 (21) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 80 (80) | 0 (0) | 6 (8) | 3 (4) | 12 (12) | 3 (3) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 10 (12) | 1 (1) | 6 (8) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 37 (37) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 (19) | 0 (0) | 16 (18) | 4 (6) | 24 (26) | 10 (10) | 10 (10) | 0 (0) | 7 (9) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 199 (200) | 0 (0) | 16 (16) | 6 (6) | 14 (15) | 8 (8) | 6 (6) | 0 (0) | 5 (5) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 13 (18) | 4 (4) | 9 (11) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 99 (100) | 0 (0) | 58 (71) | 15 (20) | 101 (127) | 41 (48) | 10 (10) | 0 (0) | 14 (16) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 116 (116) | 0 (0) | 16 (17) | 7 (9) | 26 (28) | 10 (10) | 21 (21) | 0 (0) | 11 (13) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 44 (44) | 0 (0) | 9 (9) | 3 (3) | 13 (14) | 5 (5) | 6 (6) | 0 (0) | 6 (7) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 135 (135) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 37 (66) | 5 (7) | 34 (51) | 9 (11) | 0 (0) | 0 (0) | 15 (26) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0) | 9 (10) | 0 (0) | 10 (11) | 8 (10) | 4 (4) | 0 (0) | 5 (11) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0) | 17 (17) | 6 (6) | 10 (12) | 5 (7) | 6 (6) | 0 (0) | 4 (4) | 1 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 4 (4) | 0 (0) | 9 (10) | 2 (2) | 7 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 9 (11) | 5 (12) | 4 (6) | 10 (14) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 9 (9) | 0 (0) | 2 (2) | 1 (1) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 43 (44) | 0 (0) | 37 (65) | 16 (33) | 37 (68) | 34 (55) | 12 (12) | 1 (1) | 19 (32) | 9 (25)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IVth nerve disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 6 (6) | 4 (4) | 10 (10) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Meningismus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 0 (0) | 6 (6) | 1 (1) | 12 (13) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 3 (3) | 0 (0) | 6 (7) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 4 (5) | 4 (6)
Peripheral motor neuropathy (Nervous system disorders) | 87 (87) | 0 (0) | 116 (335) | 45 (129) | 106 (273) | 57 (148) | 8 (8) | 1 (1) | 31 (72) | 23 (41)
Peripheral sensory neuropathy (Nervous system disorders) | 181 (183) | 0 (0) | 106 (273) | 41 (118) | 91 (262) | 46 (132) | 38 (38) | 0 (0) | 33 (98) | 20 (60)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 31 (32) | 0 (0) | 12 (20) | 2 (2) | 19 (20) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 3 (4)
Somnolence (Nervous system disorders) | 6 (6) | 0 (0) | 4 (4) | 8 (8) | 10 (10) | 11 (12) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 7 (8) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0) | 5 (7) | 5 (6) | 3 (3) | 6 (6) | 2 (3) | 0 (0) | 1 (2) | 2 (2)
Trigeminal nerve disorder (Nervous system disorders) | 6 (6) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 4 (4) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 8 (8) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 0 (0) | 7 (8) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Euphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 24 (24) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 0 (0) | 11 (12) | 3 (3) | 12 (12) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 1 (2) | 10 (10) | 0 (0) | 5 (5) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 6 (6) | 2 (3) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 2 (4) | 1 (1) | 9 (9) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (4) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 62 (62) | 0 (0) | 4 (14) | 1 (1) | 10 (11) | 3 (4) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 20 (20) | 0 (0) | 14 (14) | 4 (4) | 10 (11) | 6 (6) | 2 (2) | 0 (0) | 10 (10) | 6 (7)
Thromboembolic event (Vascular disorders) | 25 (25) | 0 (0) | 7 (7) | 1 (1) | 3 (3) | 3 (3) | 16 (16) | 0 (0) | 6 (6) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT00408005/Prot_SAP_000.pdf